CLINICAL TRIAL: NCT04341259
Title: A Phase I Study Of The Pharmacokinetics And Safety Of Ipatasertib In Chinese Patients With Locally Advanced Or Metastatic Solid Tumors.
Brief Title: A Study Of The Pharmacokinetics And Safety Of Ipatasertib In Chinese Participants With Locally Advanced Or Metastatic Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YP40057
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Solid Tumors
MeSH Terms: interventions — ipatasertib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ipatasertib as a Single Agent (Experimental): Participants will receive a 400-mg Ipatasertib dose (two 200-mg tablets) orally (PO) daily (QD). This study has three study periods: a screening period (up to 14 days in length), followed by a treatment period of up to approximately 2 years (Cycle 1 will be 35 days in length, all subsequent cycles will be 28 days in length) and a 28-day follow-up period after the treatment discontinuation or study completion.
  Interventions: Drug: Ipatasertib

INTERVENTIONS:
Drug: Ipatasertib — Participants will receive a 400-mg Ipatasertib dose (two 200-mg tablets) orally (PO) daily (QD) as described above.

SUMMARY:
A Phase I, Open-Label study designed to assess the pharmacokinetics (PK), safety and tolerability of ipatasertib in Chinese participants. Approximately 20 Chinese participants (12 PK-evaluable participants) with locally advanced or metastatic solid tumors for whom standard therapy either does not exist or has proven ineffective will be enrolled to provide sufficient data. Participants will receive a 400-mg ipatasertib dose (two 200-mg tablets) daily orally (PO). Participants deriving clinical benefit may be offered continued treatment with ipatasertib until disease progression, at the discretion of the investigator (as assessed by the investigator) or until the study is terminated by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented locally advanced or metastatic solid tumor that has progressed or failed to respond to at least one prior regimen.
* Not a candidate for regimens known to provide clinical benefit.
* Evaluable or measurable disease according to RECIST, v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening.
* Life expectancy of >= 12 weeks.
* Adequate haematologic and organ function within 14 days prior to initiation of study treatment.
* Women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating eggs.
* Men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm.
* Participants must reside in the People's Republic of China

Exclusion Criteria:

* Leptomeningeal disease as the only manifestation of the current tumor.
* Type 1 or 2 diabetes mellitus requiring insulin at study entry.
* Inability or unwillingness to swallow pills.
* Malabsorption syndrome or other condition that would interfere with enteral absorption.
* Known and untreated, or active CNS metastases (progressing or requiring anticonvulsants for symptomatic control).
* Congenital long QT syndrome or corrected QT interval (QTc) > 480 ms.
* Active congestive heart failure or ventricular arrhythmia requiring medication.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring weekly paracentesis for 3 consecutive weeks prior to initiation of ipatasertib treatment.
* Severe infections within 4 weeks prior to screening including but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Requirement for any daily supplemental oxygen.
* History of Inflammatory bowel disease or active bowel inflammation.
* Symptomatic hypercalcemia requiring continued use of bisphosphonate or denosumab therapy.
* Clinically significant history of liver disease, including viral disease or hepatitis,current alcohol abuse or cirrhosis.
* Known HIV infection.
* Active (chronic or acute) hepatitis C virus (HCV) at screening.
* Hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test or a positive quantitative HBV DNA test at screening
* Significant traumatic injury within 3 weeks prior to initiation of ipatasertib treatment.
* Major surgical procedure within 4 weeks prior to initiation of ipatasertib treatment.
* Treatment with chemotherapy, immunotherapy, or biologic therapy as cancer therapy within 3 weeks prior to initiation of ipatasertib treatment.
* Use of strong CYP3A4 inhibitors within 4 weeks prior to initiation of ipatasertib treatment.
* Oral endocrine therapy within 2 weeks prior to initiation of ipatasertib treatment.
* Prior treatment with a PI3-kinase inhibitor in which the patient experienced a Grade >= 3 drug-related adverse event or otherwise would be at increased risk for additional PI3K-related toxicity.
* Palliative radiation to bony metastases within 2 weeks prior to initiation of ipatasertib treatment.
* Radiotherapy (other than palliative radiation to bony metastases) as cancer therapy within 4 weeks prior to initiation of ipatasertib treatment.
* Treatment with an investigational agent within 4 weeks prior to initiation of ipatasertib treatment.
* Unresolved toxicity from prior therapy, except for alopecia and Grade 1 peripheral neuropathy.
* Pregnant or lactating.
* Inability to comply with study and follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
AUC (0-inf) after a single dose and AUC (0-24) after single and multiple doses of Ipatasertib | Up to 25 months
Maximum plasma concentration (Cmax) of Ipatasertib | Up to 25 months
Minimum plasma concentration (Cmin) of Ipatasertib after multiple doses of Ipatasertib | Up to 25 months
Time to maximum plasma concentration (tmax) of Ipatasertib | Up to 25 months
Terminal half-life (t1/2) of Ipatasertib and GO37220 | Up to 25 months
Apparent clearance (CL/F) of Ipatasertib and GO37220 after single and multiple doses of Ipatasertib | Up to 25 months
Accumulation ratio at steady state (Rcmax) of Ipatasertib | Up to 25 months
  Accumulation ratio will be calculated as follows: Rcmax = AUC24h,ss/AUC0-24 of Day 1.

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 25 months
  Assessed by the NCI CTCAE v5.0 criteria.
Percentage of Participants with Adverse Events leading to Study Treatment Discontinuation, Modification or Interruption | Up to 25 months
Number of Deaths | Up to 25 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Zhang J, Liu R, Sutaria D, Sane R, Fan M, Wang R, Song G, Chen K, Arzumanova K, Hu X. A Phase I Study of the Pharmacokinetics and Safety of Ipatasertib, an Akt Inhibitor in Chinese Patients With Locally Advanced or Metastatic Solid Tumors. Clin Ther. 2025 Feb;47(2):128-134. doi: 10.1016/j.clinthera.2024.11.021. Epub 2024 Dec 24. PMID 39721851